CLINICAL TRIAL: NCT04003961
Title: The Impact of High Risk for OSA in Prognosis and Treatment Outcomes of Lung Cancer
Brief Title: Impact of Risk for OSA in Lung Cancer
Status: Completed | Type: Observational
Sponsor: Atatürk Chest Diseases and Chest Surgery Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Sezgi Şahin Duyar, Principal Investigator, Atatürk Chest Diseases and Chest Surgery Training and Research Hospital
Other Study IDs: 1905
Record Dates: First submitted 2019-06-21; First posted 2019-07-01 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2022-01

CONDITIONS: Obstructive Sleep Apnea; Lung Cancer
Keywords: Lung Cancer; Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive; Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Moderate/high risk for OSA with EDS: All clinical data of the patients who has moderate/high risk for OSA with excessive daytime sleepiness (EDS) will be assessed with statistical methods.
  Interventions: Other: STOP- BANG Questionnaire and Epworth sleepiness scale
- Moderate/high risk for OSA without EDS: All clinical data of the patients who has moderate/high risk for OSA without excessive daytime sleepiness(EDS) will be assessed with statistical methods.
  Interventions: Other: STOP- BANG Questionnaire and Epworth sleepiness scale
- Low risk for OSA: All clinical data of the patients who has low risk for OSA will be assessed with statistical methods.
  Interventions: Other: STOP- BANG Questionnaire and Epworth sleepiness scale

INTERVENTIONS:
Other: STOP- BANG Questionnaire and Epworth sleepiness scale — STOP- BANG Questionnaire and Epworth sleepiness scale will be filled in maximum 10 minutes

SUMMARY:
Background: Previous studies have reported that intermittent hypoxia in obstructive sleep apnea (OSA) is associated with tumor progression, metastasis and treatment outcomes. However, studies explaining the relationships between specific types of cancer and OSA are needed. In this study, it is aimed to show the effect of excessive daytime sleepiness as determined by Epworth sleepiness scale(ESS) and the effect of OSA risk determined by STOP BANG questionnaire on survival and treatment outcomes in lung cancer.

Method: The patients who admit the palliative care outpatient clinic of our hospital with the diagnosis of lung cancer (stage 3 and stage 4 non-small cell lung cancer or limited / extensive stage small cell lung cancer) between July 2019-2020 will be assessed for excessive daytime sleepiness(EDS) and risk of obstructive sleep apnea (OSA) by Epworth sleepiness scale and the STOP-BANG questionnaire. The patients will be grouped according to the risk of OSA and EDS.Total / progression-free survival, treatment outcomes and side effects of the treatment will be evaluated comparatively.

DETAILED DESCRIPTION:
The patients who admit the palliative care outpatient clinic of our hospital with the diagnosis of lung cancer (stage 3 and stage 4 non-small cell lung cancer or limited / extensive stage small cell lung cancer) between July 2019-2020 prior to the treatment and the patient who has not yet completed the first-line chemotherapy with a weight loss <10% will be invited to fill the Epworth sleepiness scale and the STOP-BANG questionnaire. Patients' anthropometric measurements (height, weight, BMI, fat-free BMI, neck circumference) will be taken. The treatment outcomes and side-effects in patients with EDS and moderate / high risk for OSA will be compared with patients with low OSA risk. Demographic information (age, gender, smoking history), anthropometric measurements (height, weight, body mass index, fat free body mass index, neck circumference), clinical information (snoring, witnessed apnea, daytime excessive sleep presence of symptoms of symptoms, pulmonary function tests, radiological TNM stages, diagnostic method, diagnosis date, fiberoptic bronchoscopy findings, ECOG performance status, treatment results, treatment-related side effects) laboratory values (complete blood count results albumin, lactate dehydrogenase level) and the results of Epworth sleepiness scale and of STOP-BANG questionnaire will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18-75 years of age with the diagnosis of lung cancer (stage 3 and 4 non-small cell lung cancer or limited / extensive small cell lung cancer) and who sign the informed consent to participate in the study

Exclusion Criteria:

* Patients older than 75 years old amd younger than 18 years old
* Sedatives / anxiolytic drug users
* Neurological or psychiatric disorders
* Those who have contradictions for standard chemoradiotherapy (ECOG performance status 3-4)
* Stage 1 or stage 2 non-small cell lung cancer patients who may be referred to thoracic surgery
* Patients with brain metastasis
* People who have a shift work
* Vena cava superior syndrome
* Alcohol dependence
* Malignant airway stenosis
* Congestive heart failure (EF <50%)
* Patients with chronic renal failure

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients will be selected from the palliative care outpatient clinic according to the overmentioned criteria
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
STOP-BANG questionnaire | Up to 4 months from the initial diagnosis of lung cancer (the patients who has not initiated or has not finished the first line therapy )
  OSA - Low Risk : Yes to 0 - 2 questions OSA - Intermediate Risk : Yes to 3 - 4 questions OSA - High Risk : Yes to 5 - 8 questions or Yes to 2 or more of 4 STOP questions + male gender or Yes to 2 or more of 4 STOP questions + BMI > 35kg/m2 or Yes to 2 or more of 4 STOP questions + neck circumference 17 inches / 43cm in male or 16 inches / 41cm in female
Epworth Sleepiness Scale (ESS) | Up to 4 months from the initial diagnosis of lung cancer (the patients who has not initiated or has not finished the first line therapy will be assessed with Epworth Sleepiness Scale)
  Epworth Sleepiness Scale (ESS) is a self-administered questionnaire with 8 questions by which daytime sleepiness in eight different activities is assessed on a 4-point scale (0-3). The ESS score can range from 0 to 24. The higher the ESS score, the higher that person's 'daytime sleepiness'. ESS score ≥ 10 will be used to indicate excessive daytime sleepiness.

CONTACTS AND LOCATIONS:
Overall Officials: Sezgi Şahin Duyar, MD, Study Director — Atatürk Chest Diseases and Thoracic Surgery Traininig and Research Hospital
Locations (1):
- Atatürk Chest Diseases and Chest Surgery Training and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No